CLINICAL TRIAL: NCT05617898
Title: Determining the Role of Social Reward Learning in Social Anhedonia in First-Episode Psychosis Using Motivational Interviewing in a Perturbation-Based Neuroimaging Approach
Brief Title: Determining the Role of Social Reward Learning in Social Anhedonia
Acronym: SAMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Junghee Lee, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-300009711; 1R01MH129351-01A1 (NIH)
Record Dates: First submitted 2022-10-31; First posted 2022-11-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Psychosis
Keywords: social anhedonia, social reward learning, fMRI, sensitivity to reward
MeSH Terms: conditions — Psychotic Disorders; Anhedonia | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational Interview Intervention (Experimental): This arm involves three 45-minute sessions on motivational interviewing targeting sensitivity to social reward.
  Interventions: Behavioral: Motivational Interviewing
- Active Control Intervention (Active Comparator): This arm involves three 45-minute sessions on didactic training on nutrition.
  Interventions: Behavioral: Nutrition Didactic Training

INTERVENTIONS:
Behavioral: Motivational Interviewing — Three motivational interviewing sessions will target sensitivity to social reward, including subjective evaluation of social interaction, socially rewarding stimuli, and events (e.g., interactions with others, feedback from others).
  Arms: Motivational Interview Intervention
Behavioral: Nutrition Didactic Training — The Nutrition didactic training will ask participants to discuss pros and cons of healthy eating habits and how to improve their current eating habits.
  Arms: Active Control Intervention

SUMMARY:
This is a clinical trial study that aims to evaluate the specificity of the relationship between reduced sensitivity to social reward and social anhedonia at both behavioral and neural levels. Individuals who recently experienced their first-episode psychosis will be recruited. Participants will be randomized 1:1 to motivational interviewing or a time- and format-matched control probe. At pre- and post-probe, participants will perform two social reward learning tasks in the scanner. With this design feature, we will examine the relationship between sensitivity to social reward and reduced subjective experience of social pleasure at both the behavioral and neural levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* A first episode of a psychotic illness that began within the past three years
* Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 diagnosis of schizophrenia, schizophreniform, or schizoaffective disorder
* Taking 2nd generation antipsychotic medications
* Estimated premorbid IQ not less than 70 as assessed with the Wechsler Test of Adult Reading
* Appropriate for scanning (i.e., no pacemaker or metal implants) and expressed willingness to participate in scanning
* Sufficient fluency in English to comprehend testing procedures
* Corrected vision of at least 20/30

Exclusion Criteria:

* No evidence that substance use makes the diagnosis ambiguous (rule out substance-induced psychosis)
* No evidence of moderate or severe alcohol or substance use disorder in the past 3 months
* No clinically significant disease based on medical history (e.g., epilepsy) or significant head injury
* For females: no current pregnancy
* No sedatives or anxiolytics on the day of assessment
* No medication change 3 weeks prior to enrollment

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Response Bias | 3 weeks
  Response bias is defined as the likelihood of making one response, such as the frequently rewarded stimulus, more than the other response during the perceptual social reward learning task
the number of optimal response | 3 weeks
  The number of optimal response is defined as the number of responses choosing a stimuli with optimal outcomes (e.g., choosing a good over a neutral machine or choosing a neutral over a bad machine) during the inductive social reward learning task.
fMRI activation levels | 3 weeks
  fMRI activation is defined as beta weights from general linear model from key regions of interests including the ventromedial prefrontal cortex, dorsal anterior cingulate cortex and ventral striatum during the perceptual social reward learning task and the inductive social reward learning task.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California